CLINICAL TRIAL: NCT03780803
Title: Evaluation of Influence of Home Physical Training Program and Respiratory Rehabilitation on Quality of Life, Body Composition, and Function of Respiratory Muscles in Patients With Primary PAH, HFREF and IHD
Brief Title: Effect of Home Rehabilitation on State of Patients With PAH, HFREF and IHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N/ST/MN/16/002/1153
Record Dates: First submitted 2018-09-13; First posted 2018-12-19 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Hypertension; Heart Failure With Reduced Ejection Fraction; Ischemic Heart Disease
Keywords: cardiac rehabilitation; pulmonary rehabilitation
MeSH Terms: conditions — Hypertension, Pulmonary; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with PAH (Experimental): home cardiac rehabilitation and respiratory rehabilitation
  Interventions: Other: home cardiac rehabilitation and respiratory rehabilitation
- Patients with HFREF (Experimental): home cardiac rehabilitation and respiratory rehabilitation
  Interventions: Other: home cardiac rehabilitation and respiratory rehabilitation
- Patients with IHD (Experimental): home cardiac rehabilitation and respiratory rehabilitation
  Interventions: Other: home cardiac rehabilitation and respiratory rehabilitation
- Control group (No Intervention): No rehabilitation

INTERVENTIONS:
Other: home cardiac rehabilitation and respiratory rehabilitation
  Arms: Patients with HFREF; Patients with IHD; Patients with PAH

SUMMARY:
The aim of the study is to evaluate the influence of physical training and respiratory rehabilitation performed by patients at home on quality of life, symptoms, physical endurance, force of respiratory and skeletal muscles and body mass composition in patients with pulmonary arterial hypertension (PAH) or left ventricular heart failure with reduced ejection fraction - HFREF), or ischemic heart disease and evaluation the number of stem cells, natural lymphoid cells and distribution of subpopulations of monocytes (including proangiogenic monocytes) in examined persons and evaluation of theirs eventual influence of the course of disease.

DETAILED DESCRIPTION:
The study will be conducted on total group of 100 participants, from which 75 will be the patients with PAH (pulmonary arterial hypertension), HF-REF (heart failure with reduced ejection fraction) or IHD (ischemic heart disease).

In all participants medical anamnesis, physical examination, anthropometric measures, 6-minute walking distance (6MWD six minute walking distance) will be performed and initial functional class according WHO (World Health Organisation)/NYHA (New York Health Association)/CCS (Canadian Cardiovascular Society) classification will be evaluated. Medical history will consist of questions regarding coexisting diseases, treatment, lifestyle, family burden, etc. Quality of life will be assessed with use of The Short Form (36) Health Survey - SF-36) and Fatigue Severity Scale - FSS. Biochemical measures will be performed including, among others. brain natriuretic peptide (BNP), blood morphology, P-selectin, concentrations of cytokines such as : Interleukin 6 (IL-6), soluble Interleukin 6 receptor (sIL-6R), stromal derived factor-1 (SDF-1, CXCL12) and soluble tumor necrosis factor-like weak inducer of apoptosis (sTWEAK).

Among lab parameters routinely measured in groups of patients with PAH, HFREF, IHD performed in Cardiology Department of University Clinical Hospital during hospitalization will be used: creatinine level, uric acid level, total cholesterol, LDL (low density lipoprotein), HDL (high density lipoprotein), triglycerides levels, troponin I level, CRP (C reactive protein), BNP (brain natriuretic peptide), fasting glucose, TSH (thyroid stimulating hormone), blood morphology and arterial geometry. Fasting venous blood will be collected in 4 tubes each a 10 ml. Two tubes a 10ml (one dedicated to obtain serum ("on clot"), second with heparin) to perform biochemical analyses, tube a 10ml with EDTA (ethylenediaminetetraacetic acid) will be used to evaluate PBMC (peripheral blood mononuclear cell) (density gradient centrifugation), tube a 10ml with citrate will be used to obtain platelet lysate.

Additionally fasting venous blood will be obtained - 2 tubes a 10ml in order to assess number of stem cells, natural lymphoid cells, and distribution of subpopulations of lymphocytes.

In clinical evaluation measurement of respiratory (inspiratory and expiratory) muscles force with use of device MicroRPM (respiratory pressure meter), analysis of body mass composition with special regard to muscular mass with use of bioelectrical impedance analysis method (BIA) (Maltron) and measurement of hand grip strength with use of hand dynamometer will be performed.

During first visit also ECG (electrocardiogram) and echocardiography will be done.

The safe protocol of home physical training and respiratory rehabilitation adjusted to the clinical state of patients will be developed in the form of brochure with photos and precise description of exercises and the diary of self-control of patient in order to collect data regarding daily physical activity will be given to participants. Patients willing to take part in stage of exercises (circa 45 persons) will be trained in Rehabilitation Department how to perform exercises at homes. Easy to use devices dedicated to respiratory exercises (Pulmogain Respitrain) enabling respiratory muscles training with various degree of intensity and pedometers to assess daily motor activity will be given to patients.

Stage of exercises during which the next series of tests will be performed will last 6 months. Exercising patients will come to Rehabilitation Department on first and third month after start of rehabilitation in order to control the correctness of training performance, filling self-control diary assessment of patients compliance and eventual corrections of training program. Patients will be also under continuous phone supervision (minimally once a week) and in the case of doubts and need for consultation. After finishing exercises stage and performed clinical evaluation, patients will by themselves decide if they are willing to continue rehabilitation (will have possibility of further use of physiotherapists care), and follow up assessment will take place after 6 months from finishing exercises stage.

Comparative group will consist of patients with PAH, HF-REF, IHD who agreed to participate in study but were not qualified to the exercises stage. Control group will consist of patients of Cardiology Department and Cardiology Outpatient Clinic and Rehabilitation Department (without cardiovascular diseases). Range of examinations in control group will consists of medical anamnesis, physical examination, anthropometric measures, individually filled questionnaires SF-36 and FSS, evaluation of respiratory muscles force, hand grip strength and analysis of body mass composition BIA.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* informed consent signed by patient to conduct the study
* no diseases excluding rehabilitation
* pts with idiopathic, inherited PAH (pulmonary arterial hypertension), or in the course of connective tissue diseases, portal hypertension, congenital heart diseases.
* PAH confirmed in catheterisation of right side of heart mPAP (mean pulmonary arterial pressure) ≥25 mmHg, PCWP (pulmonary capillary wedge pressure) ≤15mmHg.
* Chronic heart failure - left ventricle ejection fraction <40% in echocardiography, NYHA *New York Health Association) class II-III
* stable ischaemic heart disease in CCS (Canadian Cardiovascular Society) class II-III

Exclusion Criteria:

* Other types of pulmonary hypertension
* COPD (chronic obstructive pulmonary disease), asthma
* malignancies
* Acute inflammatory state up to 4 weeks before inclusion to the study
* Acute coronary syndrome up to 3 months before inclusion to the study
* Heart failure in NYHA IV class
* severe anaemia (Hgb <11g/dl for men <10g/dl for women)
* electrolyte and hormonal disturbances in period of 1 month before inclusion to the study
* substantial modification of treatment of main disease within last 3 months
* ischaemic heart disease in CCS class IV
* Other clinical situations excluding to perform controlled program of rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical improvement assesment of 6 MWT distance | 6 months
  6-min walk test (6 MWT) is a exercise test that entails measurement of distance walked over a span of 6 minutes by patient good outcome > 500 m, bad outcome < 200 m

SECONDARY OUTCOMES:
Evaluation of quality of life | 6 months
  Quality of life measurement with SF36 (The Short Form (36) Health Survey, which is a 36-item, patient-reported survey of patient health.The Optum™ SF-36v2® Health Survey asks 36 questions to measure functional health and well-being from the patient's point of view. It is a practical, reliable and valid measure of physical and mental health that can be completed in five to ten minutes. The more number of points witness of better quality of life.
  Scores are calibrated so that 50 is the average score or norm. This norm-based score allows comparison among the three surveys and across the more than 19,000 studies published in the past 20 years. This bibliography includes studies of hundreds of diseases, conditions and populations, and greatly enhances the ability to interpret SF health survey data in new studies.
Force of respiratory muscles | 6 months
  measurement of maximal inspiratory and expiratory pressure
Clinical improvement - evaluation of WHO class | 6 months
  Patients' functional status is assessed with use of World Health Organisation (WHO) for pulmonary arterial hypertension. Best status is class I, worst status is class IV
Evaluation of NYHA class | 6 months
  Patients' functional status is assessed with use of New York Heart Association (NYHA) classification for heart failure, best status is class I, worst status is class IV.
Evaluation of CCS class | 6 months
  Patients' functional status is assessed with use of Canadian Cardiovascular Society (CCS) classification for coronary artery disease. Best status is class I, worst status is class IV

OTHER OUTCOMES:
Body mass composition in patients with PAH | 6 months
  Bioelectrical impedance analysis of body mass composition- body fat (amount of body fat in kilograms), body fat (amount of body fat percentage), body muscle content (amount of body muscles in kilograms), body muscle content (amount of body muscles percentage), water content (amount of water in kilograms), water content (amount of water percentage), organic substances content (amount of organic substances in kilograms), organic substances content (amount of organic substances percentage).
Weight | 6 months
  measurement of weight in kilograms
Concentration of BNP (brain natriuretic peptide) | 6 months
  Biochemical analyses - serum concentrations of brain natriuretic peptide (BNP) pg/ml
Concentration of creatinine | 6 months
  Measurement of serum concentrations of creatinine mg/dl
Concentration of uric acid | 6 months
  Measurement of serum concentrations of uric acid mg/dl
Concentration of total cholesterol | 6 months
  Measurement of serum concentrations of total cholesterol mg/dl
Concentration of LDL | 6 months
  Measurement of serum concentrations of LDL (low density lipoprotein) mg/dl
Concentration of HDL | 6 months
  Measurement of serum concentrations of HDL (high density lipoprotein) mg/dl
Concentration of triglycerides | 6 months
  Measurement of serum concentrations of triglycerides mg/dl
Concentration of CRP | 6 months
  Measurement of serum concentrations of CRP (C-reactive protein) mg/dl
Concentration of fasting glucose | 6 months
  Measurement of serum concentrations of fasting glucose mg/dl
Activity of TSH | 6 months
  Measurement of serum activity of TSH mU/l,
Concentration of Troponin I | 6 months
  Measurement of serum concentrations of troponin I µg/l,
Number of WBC | 6 months
  Measurement of number of WBC (white blood cells) K/µl,
Number of RBC | 6 months
  Measurement of number of RBC (red blood cells ) M/µl
Concentration of Hemoglobin | 6 months
  Measurement of serum concentrations of Hgb (hemoglobin) g/dl
Concentration of P selectin | 6 months
  Measurement of serum concentrations of P selectin, ng/ml
Concentration of Il-6 | 6 months
  Measurement of serum concentrations of interleukin 6 (IL-6) pg/ml
Concentration of sIl-6 R | 6 months
  Measurement of serum concentrations of soluble Interleukin 6 receptor (sIL-6R),ng/ml
Concentration of SDF-1 | 6 months
  Measurement of serum concentrations of stromal derived factor-1 (SDF-1, CXCL12), ng/ml
Concentration of sTWEAK | 6 months
  Measurement of serum concentrations of soluble tumor necrosis factor-like weak inducer of apoptosis (sTWEAK). pg/ml
Percentage of stem cells | 6 months
  assesment of amount of stem cells (percentage of undifferentiated cells)
percentage of subpopulations of monocytes | 6 months
  profile of subpopulations of monocytes (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Karol Kamiński, Professor, Study Chair — Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Department of Rehabilitation, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris NR, Kermeen FD, Holland AE. Exercise-based rehabilitation programmes for pulmonary hypertension. Cochrane Database Syst Rev. 2017 Jan 19;1(1):CD011285. doi: 10.1002/14651858.CD011285.pub2. PMID 28099988
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Background] Zafrir B. Exercise training and rehabilitation in pulmonary arterial hypertension: rationale and current data evaluation. J Cardiopulm Rehabil Prev. 2013 Sep-Oct;33(5):263-73. doi: 10.1097/HCR.0b013e3182a0299a. PMID 23962982
- [Background] Taylor RS, Sagar VA, Davies EJ, Briscoe S, Coats AJ, Dalal H, Lough F, Rees K, Singh S. Exercise-based rehabilitation for heart failure. Cochrane Database Syst Rev. 2014 Apr 27;2014(4):CD003331. doi: 10.1002/14651858.CD003331.pub4. PMID 24771460
- [Background] Sagar VA, Davies EJ, Briscoe S, Coats AJ, Dalal HM, Lough F, Rees K, Singh S, Taylor RS. Exercise-based rehabilitation for heart failure: systematic review and meta-analysis. Open Heart. 2015 Jan 28;2(1):e000163. doi: 10.1136/openhrt-2014-000163. eCollection 2015. PMID 25685361
- [Background] Oldridge N. Exercise-based cardiac rehabilitation in patients with coronary heart disease: meta-analysis outcomes revisited. Future Cardiol. 2012 Sep;8(5):729-51. doi: 10.2217/fca.12.34. PMID 23013125
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Derived] Wojciuk M, Ciolkiewicz M, Kuryliszyn-Moskal A, Chwiesko-Minarowska S, Sawicka E, Ptaszynska-Kopczynska K, Kaminski K. Effectiveness and safety of a simple home-based rehabilitation program in pulmonary arterial hypertension: an interventional pilot study. BMC Sports Sci Med Rehabil. 2021 Jul 28;13(1):79. doi: 10.1186/s13102-021-00315-y. PMID 34321095
- See also: Effectiveness and safety of a simple home-based rehabilitation program in pulmonary arterial hypertension: an interventional pilot study — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC8316895/